CLINICAL TRIAL: NCT03728634
Title: This Was a Phase 1/2, Double-blind, Randomized, Placebo-controlled, Dose-escalation Study Conducted at a Single Center for the Healthy Volunteer Cohorts in up to 56 Participants. It Consisted of 1 Single-dose Cohort and 3 Multiple-dose Cohorts (n = 12 Per Cohort, 10 Active:2 Placebo). The Open-label, hATTR Patient Cohort Portion of the Study Was Conducted at Multiple Centers.
Brief Title: Evaluate the Safety and Tolerability, as Well as the Pharmacokinetic and Pharmacodynamic Profiles of Single and Multiple Doses of Eplontersen Administered Subcutaneously to Healthy Volunteers and Patients With Hereditary Transthyretin-Mediated Amyloidosis (hATTR ).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION-682884-CS1
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers; hATTR Amyloidosis
MeSH Terms: interventions — eplontersen; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Multiple Dose Cohort: Placebo (Placebo Comparator): Participants received ION-682884 matching placebo, subcutaneously (SC) once every 4 weeks [Q4W] (total of 4 doses) along with daily oral supplemental doses of the recommended daily allowance (RDA) of vitamin A during the 13-week Treatment Period.
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin A
- Multiple Dose Cohort A: ION-682884 45 mg (Experimental): Participants received ION-682884, 45 milligrams (mg), SC, Q4W (total of 4 doses) along with daily oral supplemental doses of the RDA of vitamin A during the 13-week Treatment Period.
  Interventions: Drug: ION-682884; Dietary Supplement: Vitamin A
- Multiple Dose Cohort E: ION-682884 60 mg (Experimental): Participants received ION-682884, 60 mg, SC, Q4W (total of 4 doses) along with daily oral supplemental doses of the RDA of vitamin A during the 13-week Treatment Period.
  Interventions: Drug: ION-682884; Dietary Supplement: Vitamin A
- Multiple Dose Cohort B: ION-682884 90 mg (Experimental): Participants received ION-682884, 90 mg, SC, Q4W (total of 4 doses) along with daily oral supplemental doses of the RDA of vitamin A during the 13-week Treatment Period.
  Interventions: Drug: ION-682884; Dietary Supplement: Vitamin A
- Single Dose Cohort: Placebo (Placebo Comparator): Participants received single dose of ION-682884 matching placebo, SC along with daily oral supplemental doses of the RDA of vitamin A on Day 1.
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin A
- Single Dose Cohort C: ION-682884 120 mg (Experimental): Participants received single dose of ION-682884, 120 mg, SC along with daily oral supplemental doses of the RDA of vitamin A on Day 1.
  Interventions: Drug: ION-682884; Dietary Supplement: Vitamin A

INTERVENTIONS:
Drug: ION-682884 — ION-682884 administered SC
  Other Names: Eplontersen; AKCEA-TTR-LRx; IONIS-TTR-LRx
  Arms: Multiple Dose Cohort A: ION-682884 45 mg; Multiple Dose Cohort B: ION-682884 90 mg; Multiple Dose Cohort E: ION-682884 60 mg; Single Dose Cohort C: ION-682884 120 mg
Drug: Placebo — Placebo comparator calculated volume to match ION-682884 administered SC
  Arms: Multiple Dose Cohort: Placebo; Single Dose Cohort: Placebo
Dietary Supplement: Vitamin A — Oral supplement

SUMMARY:
To evaluate the safety and tolerability, as well as the pharmacokinetic and pharmacodynamic profiles of single and multiple doses of Eplontersen administered subcutaneously to healthy volunteers and patients with Hereditary Transthyretin-Mediated Amyloidosis (hATTR ).

DETAILED DESCRIPTION:
This will be a Phase 1/2, double-blind, randomized, placebo-controlled, dose-escalation study conducted at a single center for the healthy volunteer cohorts in up to 56 participants. It will consist of 1 single-dose cohort and 3 multiple-dose cohorts (n = 12 per cohort, 10 active:2 placebo). The open-label, hATTR patient cohort portion of the study will be conducted at multiple centers.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers (Cohorts A, B, C, and E)

1. Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal
2. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential, the subject or the subject's non-pregnant female partner must be using a highly effective contraceptive method
3. Weight ≥ 50 kg and BMI < 32 kg/m^2

Exclusion Criteria for Healthy Volunteers (Cohorts A, B, C, and E)

1. Clinically-significant (CS) abnormalities in medical history, screening laboratory results, physical or physical examination that would render a subject unsuitable for inclusion including abnormal safety labs
2. Drug or alcohol dependency or abuse
3. Treatment with another investigational drug, biological agent, or device within 1 month of Screening, or 5 half-lives of investigational agent, whichever is longer
4. Blood donation within 28 days
5. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the Study

Inclusion Criteria for hATTR Patients (Cohort D)

1. Aged 18 to 82 years at the time of informed consent
2. Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal
3. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential, the subject or the subject's non-pregnant female partner must be using a highly effective contraceptive method
4. Diagnosis of hereditary transthyretin-mediated polyneuropathy
5. BMI > 16 kg/m2

Exclusion Criteria for hATTR Patients (Cohort D)

1. Clinically-significant (CS) abnormalities in medical history, screening laboratory results, physical or physical examination that would render a subject unsuitable for inclusion, including but not limited to abnormal safety labs
2. Karnofsky performance status ≤ 50
3. Other causes of sensorimotor or autonomic neuropathy (e.g., autoimmune disease), including uncontrolled diabetes
4. Prior liver transplant or anticipated liver transplant within 1-yr of Screening
5. New York Heart Association (NYHA) functional classification of ≥ 3
6. Acute coronary syndrome or major surgery within 3 months of Screening
7. Other types of amyloidosis
8. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the Study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Pharma Services, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diep JK, Yu RZ, Viney NJ, Schneider E, Guo S, Henry S, Monia B, Geary R, Wang Y. Population pharmacokinetic/pharmacodynamic modelling of eplontersen, an antisense oligonucleotide in development for transthyretin amyloidosis. Br J Clin Pharmacol. 2022 Dec;88(12):5389-5398. doi: 10.1111/bcp.15468. Epub 2022 Aug 7. PMID 35869634
- [Derived] Viney NJ, Guo S, Tai LJ, Baker BF, Aghajan M, Jung SW, Yu RZ, Booten S, Murray H, Machemer T, Burel S, Murray S, Buchele G, Tsimikas S, Schneider E, Geary RS, Benson MD, Monia BP. Ligand conjugated antisense oligonucleotide for the treatment of transthyretin amyloidosis: preclinical and phase 1 data. ESC Heart Fail. 2021 Feb;8(1):652-661. doi: 10.1002/ehf2.13154. Epub 2020 Dec 7. PMID 33283485

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 participants were enrolled, of which 36 were randomized in multiple-dose cohorts and 11 in single-dose cohorts. This study consisted of a single-dose on Day 1, and 13 weeks of Post-Treatment Follow-up for participants in Cohort C and a 12-week Treatment Period followed by 13-week Post Treatment Evaluation Period for participants in Cohorts A, B, and E. Due to limited number of suitable participants with hereditary transthyretin amyloidosis (hATTR), Cohort D was never initiated.
Groups:
- Multiple Dose Cohort: Placebo: Participants received ION-682884 matching placebo, subcutaneously (SC), once every 4 weeks [Q4W] (total of 4 doses) along with daily oral supplemental doses of the recommended daily allowance (RDA) of vitamin A during the 13-week Treatment Period.
- Multiple Dose Cohort A: ION-682884 45 mg: Participants received ION-682884, 45 mg, SC, Q4W (total of 4 doses) along with daily oral supplemental doses of the RDA of vitamin A during the 13-week Treatment Period.
Period: Overall Study
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Started | 6 | 10 | 10 | 10 | 2 | 9
Completed | 6 | 10 | 10 | 10 | 2 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all randomized participants who received at least 1 injection of study drug (ION-682884 or placebo).
Groups:
- Multiple Dose Cohort: Placebo: Participants received ION-682884 matching placebo, SC, Q4W (total of 4 doses) along with daily oral supplemental doses of the RDA of vitamin A during the 13-week Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg | Total
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9 | 47
Age, Continuous [Mean (Full Range); unit: years] | 49.2 [39.0 to 57.0] | 51.6 [28.0 to 61.0] | 51.6 [23.0 to 65.0] | 51.1 [28.0 to 62.0] | 57.0 [53.0 to 61.0] | 43.4 [26.0 to 60.0] | 49.84 [23.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 4 | 2 | 1 | 20
  Male | 2 | 7 | 4 | 6 | 0 | 8 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 10 | 10 | 2 | 9 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 3 | 3 | 0 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 3 | 1 | 0 | 3 | 11
  White | 4 | 6 | 4 | 6 | 2 | 3 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the AE was considered related to the medicinal (investigational) product. An AE was to be regarded as a TEAE if it was present prior to receiving the first dose of study drug and subsequently worsened or was not present prior to receiving the first dose of study drug but subsequently appeared.
Time Frame: Up to Day 176
Population: Safety Set included all randomized participants who receive at least 1 injection of study drug (ION-682884 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9
Participants | 3 | 1 | 3 | 7 | 1 | 4

2. Primary Outcome: Percentage of Participants Using Concomitant Medications
Description: A concomitant therapy was any non-protocol-specified drug or substance (including over-the-counter [OTC] medications, herbal medications, and vitamin supplements) administered between signing of informed consent and the last study visit.
Time Frame: Up to Day 176
Population: Safety Set included all randomized participants who receive at least 1 injection of study drug (ION-682884 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9
percentage of participants | 0.0 | 0.0 | 30.0 | 0.0 | 0.0 | 22.2

3. Primary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Laboratory parameters included measurement of blood chemistry, hematology, coagulation, complement, or urinalysis parameters for the single-dose and multiple-dose cohorts. Number of participants with clinically significant values in laboratory based on Investigator's assessment are reported. Any value outside the normal range was to be flagged for the attention of the investigator was to assess whether or not a flagged value is of clinical significance.
Time Frame: Up to Day 176
Population: Safety Set included all randomized participants who receive at least 1 injection of study drug (ION-682884 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Physical examination included measurement of height and weight for body mass index (BMI) determination. Number of participants with clinically significant findings in physical examination based on Investigator's assessment are reported. Any value outside the normal range was to be flagged for the attention of the investigator was to assess whether or not a flagged value is of clinical significance.
Time Frame: Up to Day 176
Population: Safety Set included all randomized participants who receive at least 1 injection of study drug (ION-682884 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Values
Description: ECG measurements included assessment of ventricular rate (VR), PR interval, QR interval, QT interval, QT corrected using Fridericia's formula (QTcF), and QT corrected using Bazett's formula (QTcB). Number of participants with clinically significant values in electrocardiogram based on Investigator's assessment are reported. Any value outside the normal range was to be flagged for the attention of the investigator was to assess whether or not a flagged value is of clinical significance.
Time Frame: Up to Day 176
Population: Safety Set included all randomized participants who receive at least 1 injection of study drug (ION-682884 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Cmax: Maximum Observed Plasma Drug Concentration of ION-TTR-LRx
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose on Days 1 and 85
Population: Pharmacokinetic (PK) Set included all participants who were randomized, received at least 1 dose of ION-682884, and had at least 1 evaluable PK sample. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliters (µg/mL)
Arm/Group | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 10 | 10 | 10 | 9
micrograms per milliters (µg/mL)
  Day 1 | 0.143 (39.3) | 0.239 (62.6) | 0.332 (43.6) | 0.542 (65.0)
  Day 85: number analyzed (Participants) | 10 | 10 | 10 | 0
  Day 85 | 0.215 (66.1) | 0.282 (74.5) | 0.471 (69.5) |

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of ION-TTR-LRx
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose on Days 1 and 85
Population: PK Set included all participants who were randomized, received at least 1 dose of ION-682884, and had at least 1 evaluable PK sample. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 10 | 10 | 10 | 9
hours
  Day 1 | 2.01 [1.00 to 4.00] | 6.00 [3.00 to 12.0] | 2.25 [1.00 to 6.00] | 4.00 [1.00 to 8.00]
  Day 85: number analyzed (Participants) | 10 | 10 | 10 | 0
  Day 85 | 3.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 3.00 [1.00 to 8.00] |

8. Secondary Outcome: AUCt: Area Under the Plasma Concentration-Time Curve From Time Zero to Time t for ION-TTR-LRx
Time Frame: From 0 to 672 hours post-dose on Day 85 for Cohorts A, B, and E; 0 hours to extrapolation to infinity post-dose on Day 1 for Cohort C
Population: PK Set included all participants who were randomized, received at least 1 dose of ION-682884, and had at least 1 evaluable PK sample. Overall number analyzed are the number of participants with data available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliter (µg*h/mL)
Arm/Group | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 10 | 10 | 10 | 7
micrograms*hour per milliliter (µg*h/mL)
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 7
  Day 1 |  |  |  | 6.78 (20.3)
  Day 85: number analyzed (Participants) | 10 | 10 | 10 | 0
  Day 85 | 1.81 (36.3) | 2.73 (43.2) | 4.35 (43.2) |

9. Secondary Outcome: CL/F: Apparent Total Clearance of ION-TTR-LRx
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 10 | 10 | 10 | 7
liters per hour (L/h)
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 7
  Day 1 |  |  |  | 17.7 (20.3)
  Day 85: number analyzed (Participants) | 10 | 10 | 10 | 0
  Day 85 | 24.8 (36.3) | 22.0 (43.2) | 20.7 (43.2) |

10. Secondary Outcome: t1/2λz: Termination Half-Life of ION-TTR-LRx
Time Frame: Up to 92 hours; post-dose on Day 85 for Cohorts A, B, and E, and on Day 1 for Cohort C
Population: PK Set included all participants who were randomized, received at least 1 dose of ION-682884, and had at least 1 evaluable PK sample. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Median (Full Range); unit: days
Arm/Group | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 8 | 8 | 7
days
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 7
  Day 1 |  |  |  | 17.9 [12.8 to 40.7]
  Day 85: number analyzed (Participants) | 6 | 8 | 8 | 0
  Day 85 | 22.3 [10.3 to 52.7] | 30.3 [20.1 to 58.9] | 24.8 [15.2 to 45.0] |

11. Secondary Outcome: Ae0-24h: Amount of Administered Dose of ION-TTR-LRx Excreted in Urine Over a 24-Hour Period
Time Frame: From 0 to 24 hours post-dose on Days 1 and 85
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms (μg)
Arm/Group | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 10 | 10 | 10 | 9
micrograms (μg)
  Day 1 | 17.0 (54.1) | 23.5 (62.3) | 29.9 (146) | 87.4 (87.9)
  Day 85: number analyzed (Participants) | 10 | 10 | 9 | 0
  Day 85 | 40.6 (38.0) | 68.3 (57.2) | 133 (33.8) |

12. Secondary Outcome: Change From Baseline in Plasma Transthyretin (TTR) Levels Following Single and Multiple-dose Administration of ION-TTR-LRx
Time Frame: Baseline, Days 29 and 99
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 injection of study drug (ION-682884 or placebo). Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: milligrams per deciliters (mg/dL)
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9
milligrams per deciliters (mg/dL)
  Day 29 | -0.225 (2.935) | -13.40 (4.312) | -18.63 (4.933) | -19.42 (5.441) | 0.725 (1.732) | -20.06 (3.615)
  Day 99: number analyzed (Participants) | 6 | 10 | 10 | 10 | 0 | 0
  Day 99 | 0.908 (4.050) | -18.60 (2.911) | -22.02 (3.564) | -21.91 (5.175) |  |
Statistical Analysis 1: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort A: ION-682884 45 mg; Change From Baseline in Plasma TTR Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 29: 45 mg; Test type: Superiority; p < 0.001, Analysis of Variance(ANOVA)
Statistical Analysis 2: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort E: ION-682884 60 mg; Change From Baseline in Plasma TTR Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 29: 60 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort B: ION-682884 90 mg; Change From Baseline in Plasma TTR Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 29: 90 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 4: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort A: ION-682884 45 mg; Change From Baseline in Plasma TTR Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 99: 45 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 5: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort E: ION-682884 60 mg; Change From Baseline in Plasma TTR Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 99: 60 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 6: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort B: ION-682884 90 mg; Change From Baseline in Plasma TTR Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 99: 90 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 7: Comparison: Single Dose Cohort: Placebo vs Single Dose Cohort C: ION-682884 120 mg; Change From Baseline in Plasma TTR Levels Following Single-Dose Administration of ION-TTR-LRx at Day 29: 120 mg; Test type: Superiority; p = 0.036, ANOVA

13. Secondary Outcome: Change From Baseline in Plasma Retinol Binding Protein 4 (RBP4) Levels Following Single and Multiple-Dose Administration of ION-TTR-LRx
Time Frame: Baseline, Days 29 and 99
Population: FAS included all randomized participants who received at least 1 injection of study drug (ION-682884 or placebo). Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliters (µg/mL)
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 2 | 9
micrograms per milliliters (µg/mL)
  Day 29 | 69 (5404) | -19317 (8459) | -16383 (5191) | -21961 (8264) | 1786 (623) | -24765 (7020)
  Day 99: number analyzed (Participants) | 6 | 10 | 10 | 10 | 0 | 0
  Day 99 | 171 (4311) | -28693 (6132) | -20124 (3946) | -25365 (7275) |  |
Statistical Analysis 1: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort A: ION-682884 45 mg; Change From Baseline in Plasma RBP4 Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 29: 45 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort E: ION-682884 60 mg; Change From Baseline in Plasma RBP4 Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 29: 60 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort B: ION-682884 90 mg; Change From Baseline in Plasma RBP4 Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 29: 90 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 4: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort A: ION-682884 45 mg; Change From Baseline in Plasma RBP4 Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 99: 45 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 5: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort E: ION-682884 60 mg; Change From Baseline in Plasma RBP4 Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 99: 60 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 6: Comparison: Multiple Dose Cohort: Placebo vs Multiple Dose Cohort B: ION-682884 90 mg; Change From Baseline in Plasma RBP4 Levels Following Multiple-Dose Administration of ION-TTR-LRx at Day 99: 90 mg; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 7: Comparison: Single Dose Cohort: Placebo vs Single Dose Cohort C: ION-682884 120 mg; Change From Baseline in Plasma RBP4 Levels Following Single-Dose Administration of ION-TTR-LRx at Day 29: 120 mg; Test type: Superiority; p = 0.036, Wilcoxon Rank Sum Exact Test (2-sided)

14. Secondary Outcome: Percent Abundance of ION-682884 Antisense Oligonucleotide (ASO) Species (Metabolite) Following Administration of ION-682884 90 mg
Description: As prespecified in the protocol, this outcome measure was planned to be analyzed only in the Multiple Dose Cohort B: 90 mg ION-682884.
Time Frame: 2 hours post-dose on Day 85
Population: PK Set included all participants who were randomized, received at least 1 dose of ION-682884, and had at least 1 evaluable PK sample. As prespecified in the protocol, this outcome measure was planned to be analyzed in healthy participants administered with 90 mg ION-682884 Q4W for 13 weeks i.e., in the Multiple Dose Cohort B: 90 mg ION-682884.
Measure: Mean (Standard Deviation); unit: percent abundance of ION-682884 ASO
Arm/Group | Multiple Dose Cohort B: ION-682884 90 mg
Number analyzed (Participants) | 10
percent abundance of ION-682884 ASO | 99.1 (1.19)

ADVERSE EVENTS:
Time Frame: Up to Day 176
Description: Safety Set included all randomized participants who received at least 1 injection of study drug (ION-682884 or placebo).
Groups:
- Single Dose Cohort C: ION-682884 120 mg: Participants received single dose of ION-682884,120 mg, SC along with daily oral supplemental doses of the RDA of vitamin A on Day 1.
Arm/Group | Multiple Dose Cohort: Placebo | Multiple Dose Cohort A: ION-682884 45 mg | Multiple Dose Cohort E: ION-682884 60 mg | Multiple Dose Cohort B: ION-682884 90 mg | Single Dose Cohort: Placebo | Single Dose Cohort C: ION-682884 120 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10 | 0/2 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10 | 0/2 | 0/9
Other Adverse Events (participants affected / at risk) | 3/6 | 1/10 | 3/10 | 7/10 | 1/2 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multiple Dose Cohort: Placebo (N=6) | Multiple Dose Cohort A: ION-682884 45 mg (N=10) | Multiple Dose Cohort E: ION-682884 60 mg (N=10) | Multiple Dose Cohort B: ION-682884 90 mg (N=10) | Single Dose Cohort: Placebo (N=2) | Single Dose Cohort C: ION-682884 120 mg (N=9)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 4 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 4 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site paraesthesia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03728634/Prot_SAP_001.pdf